CLINICAL TRIAL: NCT07335016
Title: The Role of Follicular Flushing at Oocyte Retrieval
Acronym: FOFLOR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Eugonia IVF Unit, Athens, Greece (Other)
Responsible Party: Principal Investigator, E.M. Kolibianakis, Professor in Obstetrics and Gynecology and Assisted Reproduction, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHR-18
Record Dates: First submitted 2025-11-17; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Infertility (IVF Patients); Oocyte Retrieval for IVF
Keywords: ivf; follicular flushing; oocyte retrieval
MeSH Terms: conditions — Infertility; Long Qt Syndrome 3

STUDY DESIGN:
Intervention Model Description: This study design, where each patient undergoing IVF has one ovary randomized to follicular flushing and the contralateral ovary to simple aspiration, is classified as a parallel intervention study model with within-participant (or split-body) randomization at the organ level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Follicular flushing (Active Comparator): Follicular flushing
  Interventions: Other: follicular flushing
- Simple aspiration (Active Comparator): Simple aspiration
  Interventions: Other: Simple aspiration

INTERVENTIONS:
Other: follicular flushing — Follicular flushing in IVF is a technique used during oocyte retrieval with the aim to increase the number of oocytes retrieved. In follicular flushing, after the initial aspiration, the follicle is rinsed (flushed) with a sterile fluid using the same needle. In the first arm, follicular flushing will be performed in the left ovary.
  Arms: Follicular flushing
Other: Simple aspiration — Simple aspiration in IVF is the technique used during oocyte retrieval to retrieve the oocytes from the ovaries.
  Arms: Simple aspiration

SUMMARY:
In vitro fertilization (IVF) is the most common method of medically assisted reproduction, involving fertilization of the egg by sperm in a lab. The process includes ovarian stimulation, oocyte retrieval, fertilization and culture, and embryo transfer. The success of IVF depends mainly on female age-as age increases, ovarian reserve and oocyte quality decrease-and the number of oocytes retrieved.

This study investigates whether follicular flushing during oocyte retrieval can increase the number of mature oocytes retrieved. This randomized study will be conducted in women undergoing ovarian stimulation with recombinant Folicullar Stimulating Hormone (FSH) and Gonadotropin-Releasing Hormone (GnRH) antagonist or Progestin Primed Ovarian Stimulation (PPOS) to suppress premature Luteinizing hormone (LH) rise. Final oocyte maturation will be triggered with recombinant Human chorionic gonadotropin (hCG) or GnRH agonist.

Eligible participants will have at least one follicle ≥11 mm in each ovary. On the day of oocyte retrieval, one ovary will be randomized to undergo follicular flushing using a single-lumen needle and the other simple aspiration, using the same needle. All fertilized oocytes from both ovaries will be cultured, seperately, to the blastocyst stage.

Study outcomes are the number of oocytes and mature oocytes retrieved, the oocyte retrieval rate, the mature oocyte retrieval rate, the maturation rate, the number of fertilized oocytes, the fertilisation rate, the number of blastocytes and the blastulation rate.

Sample size of 75 patients (25 per response category: poor, normal, high) provides 82-98% power to detect clinically meaningful interaction effects (Cohen's f=0.19-0.34) between response category and technique (follicular flushing vs. simple aspiration) under conservative assumptions of 50-70% of pilot study effects, lower correlations (ρ=0.35), and increased variability (α=0.05, two-sided, 5% attrition buffer.

DETAILED DESCRIPTION:
In vitro fertilization (IVF) is the most commonly applied method of medically assisted reproduction and concerns the fertilization of the egg by the sperm in a laboratory environment. The process includes the following stages: Ovarian stimulation, oocyte retrieval, fertilization and culture in the laboratory, and finally, embryo transfer.

Achieving pregnancy and live birth depends on several factors. The most important is the woman's age, as the advanced female reproductive age reduces the ovarian reserve and increases the chromosomal abnormalities of the remaining oocytes. The other important factor is the number of oocytes retrieved.

Follicular flushing aims to increase the number of mature oocytes retrieved at oocyte retrieval. The present thesis investigates the role of follicular flushing at oocyte retrieval.

The randomized study will be conducted in women undergoing ovarian stimulation with recombinant follicle-stimulating hormone (recFSH) and suppression of the premature rise of luteinizing hormone (LH) using a gonadotropin-releasing hormone (GnRH) antagonist or Progestin Primed Ovarian Stimulation (PPOS). Induction of final oocyte maturation will be done with recombinant human chorionic gonadotropin (rec hCG) or an agonist of GnRH.

Women with at least one follicle of a mean diameter of 11 millimetres or more in each ovary will be eligible to participate in the studies.

On the day of oocyte retrieval, one ovary will be randomized to undergo follicular flushing using a single-lumen needle and the other simple aspiration, using the same needle. All fertilized oocytes from both ovaries will be cultured, seperately, to the blastocyst stage.

The outcomes are the number of oocytes and mature oocytes retrieved during oocyte retrieval, the oocyte retrieval rate, the mature oocyte retrieval rate, the maturation rate, the number of fertilized oocytes, the fertilisation rate, the number of blastocytes and the blastulation rate.

This study requires 75 patients (25 per response category: poor, normal, high responders) to rigorously evaluate whether follicular flushing with single-lumen needles produces clinically meaningful improvements in oocyte yield. We employed multiple conservative assumptions to ensure adequate power even under pessimistic scenarios.

Sample size was calculated for a mixed-design ANOVA testing the Response × Technique interaction. Our published pilot study (Lainas et al., HR, 2023, N=105) using double-lumen needles demonstrated large effects, but we conservatively assume single-lumen needles will show only 50-70% of these effects. We further assumed: (1) within-ovary correlations of ρ=0.35 (lower than pilot's 0.44-0.59), (2) standard deviations 20% higher than pilot data, and (3) 90% power requirement (vs. standard 80%).

Under these ultra-conservative assumptions (50% of pilot effects), n=25 per group provides 82% power. For more realistic scenarios (70-80% of pilot effects), power exceeds 90-98%. This sample size accommodates 5% attrition (target enrollment N=79), which is appropriate for within-ovary designs where dropout is minimal. The conservative approach ensures the study can detect meaningful clinical differences while satisfying rigorous peer review standards and protecting against optimistic assumptions about equipment transition.

ELIGIBILITY:
Inclusion Criteria:

* Ovarian stimulation with recFSH and GnRH antagonist or PPOS protocol
* Triggering final oocyte maturation with hCG or GnRH agonist
* The day of oocyte retrieval at least one follicle of mean diameter of 11mm in each ovary
* ICSI method of fertilisation.

Exclusion Criteria:

* Presence of ovarian cyst of endometriosis
* History of ovarian surgery
* Monofollicular growth
* Presence of only one ovary
* Ovary not accessible at oocyte retrieval

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-01-14 (Estimated); Primary Completion 2028-01-15 (Estimated); Study Completion 2029-01-20 (Estimated)

PRIMARY OUTCOMES:
Number of oocytes retrieved | Day 0
  Oocytes retrieved at oocyte retrieval are collected in the laboratory

SECONDARY OUTCOMES:
Number of mature oocytes retrieved | Day 0
  Maturity of oocytes retrieved is observed in the laboratory about 2 hours after oocyte retrieval
Oocyte retrieval rate | Day 0
  Oocytes retrieved per mature follicles observed at the ultrasound on the day of trigger of oocyte maturation
Mature oocyte retrieval rate | Day 0
  Mature oocytes per number of mature follicles at the trigger of oocyte maturation
Rate of mature oocytes / total number of oocytes retrieved | Day 0
  Rate of mature oocytes per total number of oocytes retrieved
Number of fertilized oocytes | Day 1
  Fertilisation is observed one day after the ICSI method
Rate of fertilized oocytes / total number of mature oocytes retrieved | Day 1
  Rate of fertilized oocytes per total number of mature oocytes retrieved
Number of blastocysts | Day 5 and Day 6
  Number of blastocysts formed from the fertilised oocytes
Rate of blastocysts/total number of fertilized oocytes | Day 5 and Day 6
  Rate of blastocysts formed per total number of fertilized oocytes

CONTACTS AND LOCATIONS:
Overall Officials: Efstratios Kolibianakis, Professor, Principal Investigator — Unit of Human Reproduction, Aristotle University of Thessaloniki
Locations (2):
- Greece (2):
  - Eugonia IVF, Athens
  - Aristotle University of Thessaloniki, Thessaloniki

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lainas GT, Lainas TG, Makris AA, Xenariou MV, Petsas GK, Kolibianakis EM. Follicular flushing increases the number of oocytes retrieved: a randomized controlled trial. Hum Reprod. 2023 Oct 3;38(10):1927-1937. doi: 10.1093/humrep/dead169. PMID 37632249